CLINICAL TRIAL: NCT01943110
Title: A Clinical Trial to Evaluate the Performance and Safety of Two Intradermal Delivery Devices.
Brief Title: Evaluation of the Performance and Safety of Two Intradermal Delivery Devices.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: SID Technologies (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HS 720
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2015-04

CONDITIONS: Injections, Intradermal
Keywords: Intradermal injections; Vaccine delivery devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Saline injection with ID adapters (Experimental): Each participant will receive six injections of 0.1 ml of sterile saline solution into the skin:
  * Upper deltoid with the side-load ID adapter
  * Upper deltoid with the AD ID adapter
  * Suprascapular (behind the shoulder) with the side-load ID adapter
  * Suprascapular with the AD ID adapter
  * Forearm with the side-load ID adapter
  * Forearm with the AD ID adapter
  Interventions: Device: ID adapter (autodisable); Device: ID adapter (side load)

INTERVENTIONS:
Device: ID adapter (autodisable) — Intradermal delivery device which fits on the end of a syringe to limit the depth and angle of needle penetration into the skin. Contains an autodisable feature to prevent reuse.
  Other Names: Autodisable intradermal adapter; AD ID adapter
Device: ID adapter (side load) — Intradermal delivery device which fits on the end of a syringe to limit the depth and angle of needle penetration into the skin.

SUMMARY:
The purpose of this study is to evaluate whether two intradermal (ID) vaccine delivery devices can safely and precisely inject liquid into the intradermal layer of the skin in three different injection locations

DETAILED DESCRIPTION:
This study is a preliminary device safety and performance evaluation in healthy adult volunteers (ages 18-55 years).

Each participant will receive six injections of 0.1 ml of sterile saline solution into the skin:

* Upper deltoid with the side-load ID adapter
* Upper deltoid with the autodisable (AD) ID adapter
* Suprascapular (behind the shoulder) with the side-load ID adapter
* Suprascapular with the AD ID adapter
* Forearm with the side-load ID adapter
* Forearm with the AD ID adapter

Intradermal administration of each injection will be assessed:

* The liquid remaining on the surface of the skin will be blotted with absorbent paper and the amount of liquid present will be recorded.
* The formation of an intradermal wheal will be observed, and the diameter of the wheal measured using a ruler or similar measurement tool.
* A photo of the injection site will be taken.

Injections will be assessed for safety by observation of injection sites for any local adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Female and male participants ages 18 to 55 years.
* Healthy enough to participate in the clinical trial per site investigator assessment.
* Healthy skin on the upper deltoid, suprascapular, and forearm regions (both sides of the body).
* Able to provide signed informed consent and understand study procedures per ICH/GCP guidelines.
* Literate in English.
* Available by telephone 48 hours after the study visit.

Exclusion Criteria:

- Skin abnormalities on upper deltoid, suprascapular, and forearm regions of either side of the body (scars, rash, infection), tattoo at the injection site, or other skin conditions that would interfere with the ability to visualize an intradermal injection in the opinion of the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Klaff, MD, PhD, Principal Investigator — Rainier Clinical Research Center
Locations (1):
- Rainier Clinical Research Center, Renton, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline Injection With ID Adapters: Each participant will receive six injections of 0.1 ml of sterile saline solution into the skin:
  * Upper deltoid with the side-load ID adapter
  * Upper deltoid with the AD ID adapter
  * Suprascapular (behind the shoulder) with the side-load ID adapter
  * Suprascapular with the AD ID adapter
  * Forearm with the side-load ID adapter
  * Forearm with the AD ID adapter
  ID adapter (autodisable): Intradermal delivery device which fits on the end of a syringe to limit the depth and angle of needle penetration into the skin. Contains an autodisable feature to prevent reuse.
  ID adapter (side load): Intradermal delivery device which fits on the end of a syringe to limit the depth and angle of needle penetration into the skin.
Period: Overall Study
Arm/Group | Saline Injection With ID Adapters
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Healthy adults aged 18-55 years.
Arm/Group | Saline Injection With ID Adapters
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 38 [19 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Injections Delivered to the Intradermal Layer of the Skin
Description: The proportion of saline injections resulting in delivery to the intradermal layer of the skin will be assessed by measurement of intradermal wheals with diameters ≥ 5mm and the volume of liquid injected.
Time Frame: 1 day
Measure: Number; unit: Injections
Units Other Than Participants: Injections
Groups:
- ADID Deltoid: Injections given with the autodisable ID adapter in the deltoid region
- ADID Forearm: Injections given with the autodisable ID adapter in the forearm
- ADID Suprascapular: Injections given with the autodisable ID adapter in the suprascapular region
- SLA Deltoid: Injections given with the side-load ID adapter in the deltoid region
- SLA Forearm: Injections given with the side-load ID adapter in the forearm
- SLA Suprascapular: Injections given with the side-load ID adapter in the suprascapular region
Arm/Group | ADID Deltoid | ADID Forearm | ADID Suprascapular | SLA Deltoid | SLA Forearm | SLA Suprascapular
Number analyzed (Participants) | 29 | 30 | 30 | 30 | 30 | 30
Number analyzed (Injections) | 29 | 30 | 30 | 30 | 30 | 30
Injections
  Wheal diameter >=5mm | 28 | 30 | 30 | 30 | 30 | 30
  Leakage <=10% | 28 | 30 | 29 | 30 | 30 | 30

2. Secondary Outcome: Proportion of Injections With Safety Events
Description: The proportion of injections with safety events will be calculated for events occurring within 30 minutes and within 48 hours of injection.
Time Frame: Within 30 minutes and within 48 hours of injection
Measure: Number; unit: percentage of injections
Units Other Than Participants: Injections
Groups:
- AD ID Adapter: Injections given with the autodisable ID adapter
- SLA ID Adapter: Injections given with the side-load ID adapter
Arm/Group | AD ID Adapter | SLA ID Adapter
Number analyzed (Participants) | 30 | 30
Number analyzed (Injections) | 89 | 90
percentage of injections
  Local AE at 30 minutes post-injection | 5.6 | 4.4
  Local AE at 2 days post-injection | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 days
Description: Certain signs and symptoms were pre-specified in the case report form for participants in the study. These included bleeding, redness, pain, bruising, and abrasion at the injection site. There was also space for recording other local or systemic AEs.
Groups:
- ADID Forearm: Injections given with the autodisable ID adapter in the forearm region
- SLA Forearm: Injections given with the side-load ID adapter in the forearm region
Arm/Group | ADID Deltoid | ADID Forearm | ADID Suprascapular | SLA Deltoid | SLA Forearm | SLA Suprascapular
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 11/30 | 12/30 | 10/30 | 10/30 | 14/30 | 12/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADID Deltoid (N=30) | ADID Forearm (N=30) | ADID Suprascapular (N=30) | SLA Deltoid (N=30) | SLA Forearm (N=30) | SLA Suprascapular (N=30)
Local AE at injection site 30 minutes after injection (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 1 (1) — Local AEs reported included pain, redness, bruising, and abrasion. All were minor and resolved within 1 day following injections.
Abrasion at injection site immediately after injection (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Drop of blood at injection site immediately after injection (Skin and subcutaneous tissue disorders) | 10 (10) | 9 (9) | 10 (10) | 8 (8) | 13 (13) | 11 (11)
Systemic AE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local AEs at injection site 2 days after injection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor, funder, and PI of this study have jointly published the results.